CLINICAL TRIAL: NCT05685394
Title: Dapagliflozin Cardiovascular Effects on Patients at End-stage Renal Disease
Acronym: Dare-Esrd
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Full Professor of Cardiology and Chairman of the Laboratory of Atherosclerosis and Vascular Biology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: End-stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg P.O. daily for 6 months add-on to standard treatment
  Interventions: Drug: Dapagliflozin
- Control (No Intervention): No intervention. Patients will be followed for 6 months on their standard treatment.

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10mg P.O. daily
  Arms: Dapagliflozin

SUMMARY:
Treatment with sodium glucose co-transporter type 2 inhibitors (Sglt2i) reduced the incidence of cardiovascular death and hospitalization for heart failure by 29% in individuals with moderate chronic kidney disease. Recent observations found that beyond its effect on natriuresis, Sglt2i directly interacts with cardiomyocytes inducing improvement of myocardial function. This effect is not mitigated as glomerular filtration rate declines. Therefore, plausibly treatment with Sglt2i may attenuate heart failure in individuals end-stage kidney disease (ESKD) requiring dialysis, in whom cardiovascular disease remains the leading cause of death.

In this context, this project was designed to estimate the effect of dapagliflozin on myocardial function of dialysis subjects. Individuals with diagnosed ESKD on dialysis for at least 3 months, from both sexes, aged more than 18 years of age are eligible. Exclusion criteria are pregnant woman, hepatic failure, and known allergy to study medications. Eligible patients will be recruited from the Nephrology Division of the Clinics Hospital of the University of Campinas (Unicamp). The study was designed as a prospective, randomized, open-label, phase 4 clinical trial. Patients will be randomized, 1:1, for a 6-months treatment with either dapagliflozin 10mg/day (n=40) add to standard treatment or standard treatment alone (n=40). At the randomization visit, all patients will undergo a detailed interview and medical examination by the physician-researcher, echocardiogram and blood samples will be collected for further biochemical analysis and follow up visits will be scheduled every month for endpoints disclosure and medications dispensation until the end of study participation at the 6th month visit when echocardiogram and blood sample collection will be repeated.

Primary goal will be the difference between groups in mean change of NTproBNP levels during treatment. Secondary endpoints encompass the mean change in ejection fraction, e/e' ratio, global longitudinal and radial strain and indexed left ventricle mass. Changes in bone metabolsm and structure, assessed by serum levels of FGF-23 and α-Klotho, and changes in bone mineral density will be compared between groups as an exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* On regular dialysis regimen for at least 3 months

Exclusion Criteria:

* Known allergy to any of the investigational drug components
* Current use of sodium-glucose co-transporter 2 inhibitors
* Pregnant woman
* Myocardial infarction or myocardial revascularization in the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | 6 months
  Difference between groups in NT-proBNP change from baseline

SECONDARY OUTCOMES:
Echocardiography | 6 months
  Difference between groups from baseline of the following: ejection fraction, e/e' ratio, global longitudinal and radial strain and indexed left ventricle mass

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisas Clínicas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data may be shared on reasonable request.